CLINICAL TRIAL: NCT02237118
Title: Prospective, Randomized, Non-inferiority Investigation to Compare Effects of Mepitel® One and UrgoTul® Dressings in Acute Wound Management (Only)"
Acronym: Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPTO 05
Record Dates: First submitted 2014-09-05; First posted 2014-09-11 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2014-09

CONDITIONS: Pain
Keywords: Acute; wound; management; measured; Visual analoge scale
MeSH Terms: conditions — Pain; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepitel One (Active Comparator): Pain on dressing removal, by VAS
  Interventions: Device: Mepitel One; Device: UrgoTul
- UrgoTul (Active Comparator): Pain on removal by VAS
  Interventions: Device: Mepitel One; Device: UrgoTul

INTERVENTIONS:
Device: Mepitel One
Device: UrgoTul

SUMMARY:
To compare the effects of pain of the two dressings, Mepitel® One and UrgoTul® in acute wound management.

ELIGIBILITY:
Inclusion Criteria:

1. Acute wound: traumatic wound (dermabrasion, skin tears, other), benign burn requiring the use of dressings
2. Acute wound size between 3 cm² and 240 cm2 (wound could be covered by 2 investigational products maximum)
3. Wound whose duration is ≤ 3 days
4. Both gender with an age ≥ 18 years
5. Subject able to understand and voluntarily sign the informed consent
6. Subject able to follow the protocol
7. Subject insured to the French social security system

Exclusion Criteria:

1. Surgical wound
2. Infected, moderately to strongly exudative and haemorrhagic wound
3. Diagnosed underlying disease (e.g. diabetic neuropathy, stroke, …) which, as judged by the investigator, could interfere with the pain assessment
4. Known allergy/hypersensitivity to any of the components of the investigational products
5. Participation in other clinical investigation within one month prior to start of investigation
6. Pregnant or breast-feeding women
7. Person protected by a legal regime (tutorship or guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solanilla, Dr, Principal Investigator — Clinique Mutualiste du Medoc
Locations (1):
- Clinique Mutualiste du Medoc, Lespare, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepitel One: Pain on dressing removal, by VAS
  Mepitel One
- UrgoTul: Pain on removal by VAS
  UrgoTul
Period: Overall Study
Arm/Group | Mepitel One | UrgoTul
Started | 60 | 63
Completed | 59 | 62
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — consent withdrawn | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mepitel One; UrgoTul: Pain on dressing removal, by VAS
  Mepitel One
  UrgoTul
- Total: Total of all reporting groups
Arm/Group | Mepitel One | UrgoTul | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (21.2) | 59.8 (23.0) | 62.3 (22.2)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 29 | 32 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 29 | 35 | 64
Region of Enrollment [Number; unit: participants]
  France | 60 | 63 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-Painful Dressing Removal, Measured by Visual Aanalog Scale (VAS)
Description: To compare the effects of pain of the two dressings, Mepitel® One and UrgoTul®, during the first dressing removal. Pain measured by VAS Score ≥ 30 mm on the 100 mm VAS scale are reported.
Time Frame: 21 days
Population: intention to treat.Participants with None painfull dressing removal.
Measure: Number; unit: participants
Groups:
- Mepitel One; UrgoTul: Non-Painful dressing removal, measured by VAS
  Mepitel One
  UrgoTul
Arm/Group | Mepitel One | UrgoTul
Number analyzed (Participants) | 59 | 62
participants | 44 | 39

2. Secondary Outcome: Complete Healing at Day 21, Will be Measured Using PictZar ( Digital Planimetric System) System.
Description: Complete healing at day 21, will be measured using PictZar system.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: percentage of wound size reduction
Groups:
- Mepitel One: Complete healing was reported for 39 subjects ( 68,4%) in the Mepitel One group.
- UrgoTul: Complete healing was reported for 27 subjects ( 49,1%) in theUrgoTul group.
Arm/Group | Mepitel One | UrgoTul
Number analyzed (Participants) | 60 | 63
percentage of wound size reduction | 0.89 (1.97) | 0.52 (1.09)

3. Secondary Outcome: Condition of the Wound, Will be Assesst by the Investigator.
Description: wound size estimation, assesstemnt of the wound,
Time Frame: 21 days
Population: Missing value for some patients
Measure: Count of Participants; unit: Participants
Groups:
- Condition of the Wound Mepitel One: Condition of the wound assesed by the investigator
- Condition of the Wound, UrgoTul: Condition of the wound, UrgoTul, assessed by the investigator
Arm/Group | Condition of the Wound Mepitel One | Condition of the Wound, UrgoTul
Number analyzed (Participants) | 60 | 63
Participants
  Bleeding: number analyzed (Participants) | 59 | 58
  Bleeding: None | 41 | 38
  Bleeding: Mild | 16 | 18
  Bleeding: Moderate | 2 | 2
  Maceration: number analyzed (Participants) | 59 | 58
  Maceration: None | 50 | 42
  Maceration: Mild | 5 | 14
  Maceration: Moderate | 4 | 2
  Granulation tissue in growth in the dressing holes: number analyzed (Participants) | 58 | 57
  Granulation tissue in growth in the dressing holes: None | 37 | 39
  Granulation tissue in growth in the dressing holes: Mild | 12 | 13
  Granulation tissue in growth in the dressing holes: Moderate | 9 | 5

4. Secondary Outcome: Safety
Description: Adverse Event, Adverse Device Event
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Groups:
- Safety Mepitel One; Safety UrgoTul: Adverse Event and Adverse Device Effect
Arm/Group | Safety Mepitel One | Safety UrgoTul
Number analyzed (Participants) | 60 | 63
Participants
  Subject with Adverse Event | 6 | 7
  Subject with Adverse Device Effect | 1 | 0
  Subject with non AE | 53 | 56

5. Secondary Outcome: Assessment of the Surrounding Skin.
Description: assessment of the surrounding skin.
Time Frame: 21 days
Measure: Number; unit: percentage of patients
Groups:
- Mepitel One; UrgoTul: Condition of the surrounding skin
Arm/Group | Mepitel One | UrgoTul
Number analyzed (Participants) | 60 | 63
percentage of patients
  Inflammatory signs | 4 | 7
  Irritation | 2 | 3
  Allergic rash | 0 | 1
  Blistering | 1 | 1
  Skin stripping | 0 | 1
  Maceration | 1 | 0
  Dry | 1 | 2
  Trauma to wound edges | 1 | 4
  Product degradation on the skin | 0 | 1
  Hematoma | 5 | 1
  other | 1 | 2

ADVERSE EVENTS:
Groups:
- UrgoTul: Pain on removal by VAS
  Mepitel One
  UrgoTul
Arm/Group | Mepitel One | UrgoTul
Serious Adverse Events (participants affected / at risk) | 1/60 | 4/63
Other Adverse Events (participants affected / at risk) | 6/60 | 7/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepitel One (N=60) | UrgoTul (N=63)
Necrosis of left heel, diabetes (Endocrine disorders) | 0 (0) | 1 (1) — Necrosis of left heel, diabetes, leading to hospitalisation
pulmonary rhythm disorder (Cardiac disorders) | 0 (0) | 1 (1) — pulmonary rhythm disorder, leading to hospitalisation
cardiac insufficiency (Cardiac disorders) | 0 (0) | 2 (2) — cardiac insufficiency, both leading to hospitalisation
Gastro intestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — gastro intestinal bleeding, life threatening
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepitel One (N=60) | UrgoTul (N=63)
cutaneous eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0) — GASTROINTESTINAL BLEEDING
ALLERGY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — ALLERGY
acute elbow cellulite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — acute elbow cellulite
another wound surinfection with stapylococcus epidermidis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — another wond surinfection with stapylococcus epidermidis
ANKLE SPRAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — ANKLE SPRAIN
ERYSIPELE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — ERYSIPELE
NECROSE necrosis on the left heel (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — NECROSE necrosis on the left heel
RIGHT BASAL PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — RIGHT BASAL PULMONARY
Hospitalization for cardiac insufficiency (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalization for cardiac insufficiency
acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — acute bronchitis
cardiorespiratory failure (Cardiac disorders) | 0 (0) | 1 (1) — cardiorespiratory failure
fall (General disorders) | 0 (0) | 1 (1) — fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No